CLINICAL TRIAL: NCT06657066
Title: EFFECTIVENESS of PROBIOTIC AS an ADJUVANT to STANDARD THERAPY VERSUS STANDARD THERAPY ALONE in ADULTS with MODERATE to SEVERE PERSISTENT ASTHMA
Brief Title: EFFECTIVENESS of PROBIOTICS in ADULTS with MODERATE to SEVERE PERSISTENT ASTHMA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, binayak singh, MD (Postgraduate Trainee), King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6952/REG/KEMU/22MD200023
Record Dates: First submitted 2024-10-19; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Asthma Patients
Keywords: Asthma; Probiotics; Standard Therapy; adjuvant
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol; Formoterol Fumarate

STUDY DESIGN:
Intervention Model Description: Randomize Clinical Trial
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm - Group A (Experimental): Standar Therapy- Daily low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram as needed Short acting beta 2 agonist (SABA)/salbutamol 100mcg ,OR as needed low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram -Long acting Beta2 Agonist (LABA)/Formeterol 6 microgram.
  Along with Probiotics i.e Saccharomyces boulardii, available in sachet from employed in this research containing 250 mg of lyophilized saccharomyces boulardii
  Interventions: Drug: Beclomethasone 200mcg, salbutamol 100mcg , Beclomethasone 200 mcg/Formoterol 6 mcg, 250 mg of lyophilized saccharomyces boulardii
- Control arm- Group B (Placebo Comparator): Standard therapy only:
  Daily low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram as needed Short acting beta 2 agonist (SABA)/salbutamol 100mcg ,OR as needed low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram -Long acting Beta2 Agonist (LABA)/Formeterol 6 microgram
  Interventions: Drug: Control (Standard treatment)

INTERVENTIONS:
Drug: Beclomethasone 200mcg, salbutamol 100mcg , Beclomethasone 200 mcg/Formoterol 6 mcg, 250 mg of lyophilized saccharomyces boulardii — Daily low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram as needed Short acting beta 2 agonist (SABA)/salbutamol 100mcg ,OR as needed low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram -Long acting Beta2 Agonist (LABA)/Formeterol 6 microgram plus Saccharomyces boulardii, available in sachet from employed in this research containing 250 mg of lyophilized saccharomyces boulardii. It was given daily for three months
  Other Names: Group A
  Arms: Intervention arm - Group A
Drug: Control (Standard treatment) — The control arm will receive only standard treatment for asthma i.e Daily low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram as needed Short acting beta 2 agonist (SABA)/salbutamol 100mcg ,OR as needed low dose inhaled corticosteroid (ICS)/ Beclomethasone 200 microgram -Long acting Beta2 Agonist (LABA)/Formeterol 6 microgram.
  Other Names: Group B
  Arms: Control arm- Group B

SUMMARY:
The objective of this study is to compare the effectiveness of probiotic as an adjuvant to standard therapy versus standard therapy alone in adult with moderate to severe persistent asthma in terms of

1. Frequency of asthma exacerbations in terms of number of asthma attacks and severity of each episode.
2. Improvement in pulmonary function tests as recorded by an increase in FEV1 and FEV1/FVC ratio.

5. HYPOTHESIS Probiotics as an adjuvant to standard therapy is more effective as compared to the standard therapy alone in managing moderate to severe persistent bronchial asthma.

DETAILED DESCRIPTION:
Design of Study This was a Randomized controlled trial

Follow up protocol The patient was evaluated at the beginning of the study, and then again at one and three months following enrolment for a follow-up evaluation of the main and secondary outcomes.

Primary outcome To assess the frequency of exacerbations within 3 months.

Secondary outcome:

To observe improvement in

1. FEV1 and the FEV1/FVC ratio. Improvement in one step and more than 12% Improvement in FEV1 from baseline. Improvement in asthma control test. Sample Size - The calculated sample size is 74 individuals (37 in each category i.e Intervention & Control arm)

Sampling technique - Simple random sampling Sample selection Inclusion Criteria

1. Patients of both genders between the ages of 18 and 80 years.
2. Diagnosed cases of moderate to severe persistent asthma, as determined by ACT Score and FEV1/FVC ratio as per operational definition.

Exclusion Criteria

1. Patients with Mild asthma.
2. Pregnant females.
3. Patients who have taken fiber supplement or probiotics during the last four weeks.
4. Other pulmonary disorders, such as Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis (ABPA), chest wall deformities, bronchiectasis, pulmonary fibrosis, and lung cancer.
5. Asthma and chronic obstructive pulmonary disease overlap syndrome (ACOS).

ELIGIBILITY:
Inclusion Criteria

1. Patient of both genders between the ages of 18 and 80 years.
2. Diagnosed cases of moderate to severe persistent asthma, as determined by ACT Score and FEV1/FVC ratio as per operational definition.

Exclusion Criteria

1. Patients with Mild asthma.
2. Pregnant females.
3. Patients who have taken fiber supplements or probiotics during the last four weeks.
4. Other pulmonary disorders, such as Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis (ABPA), chest wall deformities, bronchiectasis, pulmonary fibrosis, and lung cancer.
5. Asthma and chronic obstructive pulmonary disease overlap syndrome (ACOS).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Frequencies of exacerbation | 3 months
  Assessment of the frequency of exacerbations within 3 months will be observed among the intervention & control grouo

SECONDARY OUTCOMES:
Improvment of FEV1 and FEV1/FVC ratio | 3 months
  To observe improvement in
  1. FEV1 and the FEV1/FVC ratio. Improvement in one step and more than 12% Improvement in FEV1 from baseline. Improvement in asthma control test.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Binayak Singh, MD, Principal Investigator — King Edward Medical University Lahore
Locations (1):
- King Edward Medical University, Neelagumbad, Anarkali, Lahore, Pakistan. Postal Code: 54000 Telephone: +92 (42) 99211145-54, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only the principal investigator, supervisor, and Institution Review Board will have access with patients data upon request

REFERENCES:
- See also: Clinical and molecular phenotypes of asthma are complex. The main phenotypes of adult asthma are characterized by eosinophil and/or neutrophil cell dominant airway inflammation that represent distinct clinical features. Upper and lower airways constitute — https://immunenetwork.org/DOIx.php?id=10.4110/in.2021.21.e19